CLINICAL TRIAL: NCT04805671
Title: A Phase 2/3 Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of ADG20 in the Treatment of Ambulatory Participants With Mild or Moderate COVID-19 (STAMP)
Brief Title: Evaluation of ADG20 for the Treatment of Mild or Moderate COVID-19
Acronym: STAMP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: All primary efficacy data has been collected and analyzed. Based on the safety data gathered to date, it has been determined that continued participation by study subjects would not yield any additional beneficial safety information.
Sponsor: Invivyd, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADG20-TRMT-001
Record Dates: First submitted 2021-03-17; First posted 2021-03-18 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ADG20; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The investigator, participant and sponsor personnel involved in study intervention and study evaluation will be unaware of the intervention assignments. Investigators will remain blinded to each participant's assigned study treatment throughout the course of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ADG20 IM (Experimental): Participants will be dosed on Day 1 with ADG20 IM
  Interventions: Drug: ADG20
- Placebo IM (Placebo Comparator): Participants will be dosed on Day 1 with placebo IM
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: ADG20 — Single dose of ADG20
  Arms: ADG20 IM
Drug: Normal saline — Single dose of normal saline
  Arms: Placebo IM

SUMMARY:
This placebo controlled study is intended to generate safety and efficacy data in order to provide a treatment option for COVID-19 in patients with a high risk of disease progression based on age or co-morbid medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Has had SARS-CoV-2 positive antigen, RT-PCR, or other locally approved molecular diagnostic assay obtained within 5 days prior to randomization
* Has had symptoms consistent with COVID-19 with onset 5 days before randomization
* Has one or more COVID-19-related signs or symptoms on the day of randomization
* Phase 2: Is an adult aged 18 years and above
* Phase 3: Is an adult aged 18 years and above or is an adolescent aged 12 to 17 years (inclusive) and weighing ≥40 kg at the time of screening

Exclusion Criteria:

* Is currently hospitalized or in the opinion of the investigator is anticipated to require hospitalization within 48 hours of randomization.
* Has severe COVID-19 or is on supplemental oxygen
* Has a history of a positive SARS-CoV-2 antibody serology test
* Has participated, within the last 30 days, in a clinical study involving an investigational intervention
* Has received a SARS-CoV-2 vaccine, monoclonal antibody, or plasma from a person who recovered from COVID-19 any time prior to participation in the study

NOTE: Other protocol defined inclusion/exclusion criteria apply

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 399 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-11-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (56):
- Argentina (6):
  - Adagio Investigative Site, Estomba, Buenos Aires
  - Adagio Investigative Site, Munro, Buenos Aires
  - Adagio Investigative Site, Río Cuarto, Córdoba Province
  - Adagio Investigative Site, Rosario, Santa Fe Province
  - Adagio Investigative Site, San Miguel de Tucumán, Tucumán Province
  - Adagio Investigative Site, Mar del Plata
- Brazil (5):
  - Adagio Investigative Site, Salvador, Estado de Bahia
  - Adagio Investigative Site, Taguatinga, Federal District
  - Adagio Investigative Site, Belo Horizonte, Minas Gerais
  - Adagio Investigative Site, Passo Fundo, Rio Grande do Sul
  - Adagio Investigative Site, São Paulo
- Bulgaria (8):
  - Adagio Investigative Site, Dupnitsa, Kyustendil
  - Adagio Investigative Site, Samokov, Sofia
  - Adagio Investigative Site, Sofia, Sofia-Grad
  - Adagio Investigative Site, Blagoevgrad
  - Adagio Investigative Site, Montana
  - Adagio Investigative Site, Pleven
  - Adagio Investigative Site, Rousse
  - Adagio Investigative Site, Stara Zagora
- Germany (4):
  - Adagio Investigative Site, Frankfurt am Main, Hesse
  - Adagio Investigative Site, Cologne, North Rhine-Westphalia
  - Adagio Investigative Site, Koblenz, Rhineland-Palatinate
  - Adagio Investigative Site, Berlin
- Greece (5):
  - Adagio Investigative Site, Pátrai, Achaïa
  - Adagio Investigative Site, Athens, Attica
  - Adagio Investigative Site, Heraklion, Crete
  - Adagio Investigative Site, Ioannina
  - Adagio Investigative Site, Nikaia
- Hungary (3):
  - Adagio Investigative Site, Szeged, Csongrád megye
  - Adagio Investigative Site, Székesfehérvár, Fejér
  - Adagio Investigative Site, Debrecen, Hajdú-Bihar
- Adagio Investigative Site, Chisinau, Moldova
- Poland (4):
  - Adagio Investigative Site, Krakow, Lesser Poland Voivodeship
  - Adagio Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Adagio Investigative Site, Lódz, Lódzkie
  - Adagio Investigative Site, Skierniewice, Lódzkie
- Adagio Investigative Site, Bucharest, București, Romania
- South Africa (13):
  - Adagio Investigative Site, Welkom, Free State
  - Adagio Investigative Site, Johannesburg, Gauteng
  - Adagio Investigative Site, Kempton Park, Gauteng
  - Adagio Investigative Site, Pretoria, Gauteng
  - Adagio Investigative Site, Tembisa, Gauteng
  - Adagio Investigative Site, Rustenburg, North West
  - Adagio Investigative Site, Three Rivers, Vereeniging
  - Adagio Investigative Site, Cape Town, Western Cape
  - Adagio Investigative Site, George, Western Cape
  - Adagio Investigative Site, Somerset West, Western Cape
  - Adagio Investigative Site, Worcester, Western Cape
  - Adagio Investigative Site, George
  - Adagio Investigative Site, Pretoria
- Ukraine (6):
  - Adagio Investigative Site, Dnipro, Dnipropetrovsk Oblast
  - Adagio Investigative Site, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Adagio Investigative Site, Kherson, Kherson Oblast
  - Adagio Investigative Site, Kharkiv
  - Adagio Investigative Site, Kiyiv
  - Adagio Investigative Site, Kyiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ison MG, Popejoy M, Evgeniev N, Tzekova M, Mahoney K, Betancourt N, Li Y, Gupta D, Narayan K, Hershberger E, Connolly LE, Yalcin I, Das AF, Genge J, Smith M, Campanaro E, Hawn P, Schmidt P; STAMP Study Group. Efficacy and Safety of Adintrevimab (ADG20) for the Treatment of High-Risk Ambulatory Patients With Mild or Moderate Coronavirus Disease 2019: Results From a Phase 2/3, Randomized, Placebo-Controlled Trial (STAMP) Conducted During Delta Predominance and Early Emergence of Omicron. Open Forum Infect Dis. 2023 May 24;10(6):ofad279. doi: 10.1093/ofid/ofad279. eCollection 2023 Jun. PMID 37351456
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADG20 IM | Placebo IM
Started | 198 | 201
Completed | 8 | 10
Not Completed | 190 | 191
Not completed — Death | 2 | 7
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 9 | 7
Not completed — Study terminated prematurely; participants active in the study discontinued from the trial. | 178 | 177

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | ADG20 IM | Placebo IM | Total
Number analyzed (Participants) | 198 | 201 | 399
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 150 | 152 | 302
  >=65 years | 47 | 49 | 96
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 55 [43 to 65] | 53 [41 to 65] | 54 [42 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 113 | 104 | 217
  Male | 85 | 97 | 182
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 198 | 199 | 397
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 17 | 31
  White | 183 | 181 | 364
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Greece | 9 | 11 | 20
  Romania | 18 | 18 | 36
  Ukraine | 36 | 36 | 72
  Brazil | 0 | 2 | 2
  Poland | 13 | 13 | 26
  South Africa | 20 | 20 | 40
  Bulgaria | 101 | 100 | 201
  Germany | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Incidence of COVID-19 Related Hospitalizations or All-cause Death
Description: To evaluate the efficacy of ADG20 compared to placebo in the treatment of mild or moderate COVID-19 in participants at high risk of disease progression. Hospitalization is defined as ≥24 hours of acute care in a hospital or acute care facility (includes emergency rooms, intensive care units, acute care facilities created for COVID-19 pandemic hospitalization needs, or other acute care facilities). All-cause death is defined as death for any reason from Day 1 (postdose) through Day 29.
Time Frame: Through Day 29
Population: Modified Full Analysis Set (mFAS-non-Omicron): All randomized participants with COVID-19 due to Whole Genome WGS)-confirmed or suspected non-Omicron SARS-CoV-2 variants.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 169 | 167
Participants | 8 | 23
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; ADG20 vs Placebo; Test type: Superiority; p = 0.0047, Regression, Logistic; Risk Difference (RD) = -8.7, 95% CI 2-sided [-14.71 to -2.67]; A statistical method described in Ge et al. (2011) was used to compute a population-level estimate for the treatment difference (in terms of difference in proportion) with adjustment for the pre-defined prognostic factors. The variance of the estimated treatment difference or relative risk reduction was estimated using the delta method

2. Primary Outcome: Incidence of Treatment-emergent Adverse Events
Description: Proportion of participants with at least one treatment emergent AE
Time Frame: Through day 29
Population: Safety Set: All participants who received any amount of study drug. Participants were analyzed based on the actual treatment (ADG20 versus Placebo) received. Participants with more than one AE were only counted once.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 192 | 200
Participants | 47 | 62

3. Primary Outcome: Incidence of Solicited Injection Site Reactions
Description: Proportion of participants with at least one solicited injection site reaction
Time Frame: Through Day 4
Population: Safety Set: All participants who received any amount of study drug. Participants were analyzed based on the actual treatment (ADG20 versus Placebo) received.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 192 | 200
Participants | 25 | 19

4. Primary Outcome: Changes From Baseline in Clinical Laboratory Tests (ie, CBC With Differential, Serum Chemistry, Coagulation)
Description: Proportion of participants with a potentially clinically significant change from baseline in post-baseline laboratory parameters - data presented for any analyte with >/= 2% in any arm
Time Frame: Through Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 192 | 200
Participants
  Lymphocytes (10^9/L) - L | 3 | 4
  Alanine Aminotransferase (U/L) - H | 6 | 10
  Albumin (g/L) - L | 0 | 5
  Creatinine (mcmol/L) - H | 26 | 23
  Creatinine Clearance, Estimated (mL/min/1.73m2) - L | 15 | 18
  Glucose (mmol/L) - H | 12 | 16
  Sodium (mmol/L) - L | 1 | 4
  Urea Nitrogen (mmol/L) - H | 26 | 21
  Prothrombin Intl. Normalized Ratio - H | 5 | 1

5. Primary Outcome: Changes From Baseline in Vital Signs (Body Temperature, Heart Rate, Respiration Rate, and Systolic and Diastolic Blood Pressure)
Description: Participants with Potentially Clinically Significant Changes (PCS) From Baseline in Vital Signs (Body Temperature, Heart Rate, Respiration Rate, and Systolic and Diastolic Blood Pressure) at Any Time Post-Baseline
Time Frame: Through Day 29
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 192 | 200
Participants
  SBP <=90 mmHg or Decrease >=20 mmHg | 17 | 23
  SBP >=180 mmHg or Increase >=20 mmHg | 29 | 26
  DBP <=50 mmHg or Decrease >=15 mmHg | 25 | 26
  DBP >=105 mmHg or Increase >=15 mmHg | 24 | 31
  HR <=50 bpm or Decrease >=15 bpm [a] | 78 | 96
  HR >120 bpm or Increase >=15 bpm | 20 | 25
  Temp <35 C or Decrease >=1 C [b] | 60 | 56
  Temp >=38 C or Increase >=1 C [c] | 5 | 17
  RR <=8 breaths/min or Decrease >=4 bpm | 20 | 25
  RR >=30 breaths/min or Increase >=10 bpm [d] | 2 | 2
  SpO2 <=93% or Decrease >=3% | 14 | 19

6. Secondary Outcome: Incidence of COVID-19 -Related Medically Attended Visits or All-cause Death
Description: Proportion of participants with COVID-19-related medically attended visit (telemedicine, physician office, urgent care center, emergency room, hospitalization) or all-cause death through Day 29. In addition to events defined as the primary efficacy endpoint, this endpoint also includes any medically attended visits, in-person, or telemedicine, not specified in the protocol. These include unscheduled in-person or telemedicine visits conducted by the investigator for the purpose of evaluating worsening signs or symptoms attributed to COVID-19 or emergency room, urgent care center or physician office visits, or hospitalization for attention to worsening signs or symptoms attributed to COVID-19, in the opinion of the investigator. Incidence of COVID-19-related medically attended visits or all-cause death includes participants who met any event defined for this endpoint. Participants were counted only once even if multiple events were met in the time frame.
Time Frame: Through Day 29
Population: Modified Full Analysis Set (mFAS-non-Omicron): All randomized participants with COVID-19 due to Whole Genome Sequencing (WGS)-confirmed or suspected non-Omicron SARS-CoV-2 variants.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 169 | 167
Participants | 9 | 29
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; ADG20 vs Placebo; Test type: Superiority; p = 0.0007, Regression, Logistic; Risk Difference (RD) = -11.3, 95% CI 2-sided [-17.86 to -4.81]; [other analysis details as in outcome 1, analysis 1]

7. Secondary Outcome: Incidence of COVID-19 -Related Emergency Room Visits, COVID-19-related Hospitalization, or All Cause-death
Description: Proportion of participants with any COVID 19-related emergency room visits, COVID-19-related hospitalization, or all cause death through Day 29. Defined as any stay in a hospital or acute care facility regardless of duration (includes emergency rooms, intensive care units, acute care facilities created for COVID-19 pandemic hospitalization needs, or other acute care facilities) for attention to worsening signs or symptoms attributed to COVID-19 in the opinion of the investigator or all cause death through Day 29. Incidence of COVID-19-related emergency room visits, COVID-19-related hospitalization, or all-cause death includes participants who met any event defined for this endpoint. Participants were counted only once even if multiple events were met in the time frame.
Time Frame: Through Day 29
Population: Modified Full Analysis Set (mFAS-non-Omicron): All randomized participants with COVID-19 due to WGS-confirmed or suspected non-Omicron SARS-CoV-2 variants.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 169 | 167
Participants | 8 | 23
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; ADG20 vs Placebo; Test type: Superiority; p = 0.0047, Regression, Logistic; Risk Difference (RD) = -8.7, 95% CI 2-sided [-14.71 to -2.67]; [other analysis details as in outcome 1, analysis 1]

8. Secondary Outcome: Incidence of Severe/Critical COVID-19 or All Cause Death
Description: Proportion of participants with Severe/Critical COVID-19 or all-cause death through Day 29. All-cause death is defined as death for any reason (from Day 1postdose) through Day 29. Severity is based on the investigator's assessment of severity (eCRF COVID-19 Severity Assessment) per the protocol definitions. Incidence of Severe/Critical COVID-19 or all-cause death includes participants who met any event defined for this endpoint. Participants were counted only once even if multiple events were met in the time frame.
Time Frame: Through Day 29
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 169 | 167
Participants | 8 | 23
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; ADG20 vs Placebo; Test type: Superiority; p = 0.0007, Regression, Logistic; Risk Difference (RD) = -11.3, 95% CI 2-sided [-17.86 to -4.81]; [other analysis details as in outcome 1, analysis 1]

9. Secondary Outcome: Time to Sustained Recovery Defined as Sustained Improvement or Resolution of COVID-19 Symptoms
Description: Time to sustained recovery (improvement or resolution) of COVID-19 symptoms through Day 29: Defined as the time from the first dose date to the earliest date when sustained improvement or sustained resolution of COVID-19 symptoms is met (as detailed below) through Day 29. COVID-19 symptoms assessed include fever, chills, cough, sore throat, congestion, shortness of breath/difficulty breathing at rest, shortness of breath/difficulty breathing with exertion, muscle or body aches, fatigue, headache, nausea, vomiting, and diarrhea. Loss of taste/smell is excluded from this analysis.
Time Frame: Through Day 29
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 169 | 167
Days | 11 [9 to 14] | 14 [12 to 17]
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; ADG20 vs. Placebo; Test type: Superiority; p = 0.0938, Regression, Cox; Hazard Ratio (HR) = 1.237, 95% CI 2-sided [0.964 to 1.586]

10. Secondary Outcome: Incidence of All-cause Mortality
Description: Defined as death for any reason from Day 1 (postdose). In the overall survival analysis, participants who are alive or lost to follow-up at the time of analysis are censored at the date of last contact.
Time Frame: Through Day 90
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 169 | 167
Participants | 1 | 7
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; ADG20 vs Placebo; Test type: Superiority; p = 0.0361, Regression, Cox; Hazard Ratio (HR) = 0.137, 95% CI 2-sided [0.016 to 1.162]

11. Secondary Outcome: Time to Sustained Resolution of COVID-19 Symptoms as Measured in the Daily COVID-19 Symptom Diary
Description: Time to sustained resolution of COVID-19 symptoms through Day 29: Defined as time from the dose date to the first date when all of the defined symptoms are scored as absent with no symptom recurrence or new symptoms, except cough, fatigue, and headache which may be mild or absent, through Day 29.
Time Frame: Through Day 29
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 169 | 167
Days | 13 [10 to 15] | 16 [13 to 20]
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; ADG20 vs Placebo; Test type: Superiority; p = 0.0781, Regression, Cox; Hazard Ratio (HR) = 1.255, 95% CI 2-sided [0.974 to 1.617]

12. Secondary Outcome: Change From Baseline in SARS-CoV-2 Viral Load (log10 Copies/mL) to Day 7 (±1)
Description: Assessed by RT qPCR From NP (Nasopharyngeal) Samples
Time Frame: Day 7 (±1)
Population: Modified Full Analysis Set (mFAS-non-Omicron-NP): All randomized participants with COVID-19 due to Whole Genome Sequencing (WGS)-confirmed or suspected non-Omicron SARS-CoV-2 variants with a positive baseline NP sample.
Measure: Least Squares Mean (Standard Error); unit: log10 copies/mL
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 147 | 149
log10 copies/mL | -3.61 (0.238) | -3.44 (0.224)
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; ADG20 vs. Placebo; Test type: Superiority; p = 0.4976, ANCOVA; Mean Difference (Final Values) = -0.17, 95% CI 2-sided [-0.66 to 0.32]

13. Secondary Outcome: Duration of SARS-CoV-2 Shedding Assessed by RT-qPCR From Saliva Samples
Description: Duration of SARS-CoV-2 viral shedding is defined as time from the dose date to the first date the viral load is not detected, ie, below the limit of detection (LOD), and sustained through Day 29. Participants who do not have the defined event or who discontinue study prior to Day 29 are censored at the earlier date of the last viral load assessment or Day 30. Deaths occurring prior to Day 29 were censored at Day 30.
Time Frame: Through Day 29
Population: Modified Full Analysis Set (mFAS-non-Omicron-S): All randomized participants with COVID-19 due to Whole Genome Sequencing (WGS)-confirmed or suspected non-Omicron SARS-CoV-2 variants with a positive baseline saliva sample.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 147 | 149
Days | 14 [14 to 21] | 21 [14 to 21]
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; Test type: Superiority; p = 0.7239, Regression, Cox; Hazard Ratio (HR) = 1.048, 95% CI 2-sided [0.806 to 1.364]

14. Secondary Outcome: Viral Load >5 (log10 Copies/mL) Based on Nasopharyngeal Sampling at Day 7
Description: Proportion of participants with Viral load >5 (log10 copies/mL) on Day 7 assessed by RT-qPCR from NP sample.
Time Frame: on Day 7 (+/- 1 Day)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 148 | 146
Participants | 49 | 64
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; Test type: Superiority; p = 0.0364, Regression, Logistic; Risk Difference (RD) = -11.1, 95% CI 2-sided [-21.42 to -0.70]

15. Secondary Outcome: SARS-CoV-2 Viral Clearance (Days 5, 7, 11, 14, 21, and 29) Assessed by RT-qPCR From Saliva Samples (and NP Samples for Day 7)
Description: Proportions of SARS-CoV-2 viral clearance (Days 3, 5, 7, 11, 14, 21, and 29) assessed by RT-qPCR from saliva samples: In the mFAS-S, the cumulative proportion of participants with viral clearance (viral load not detected and sustained through Day 29) at Days 3, 5, 7, 11, 14, 21, and 29 will be assessed by RT-qPCR from saliva samples. Participants who have died or discontinued study prior to Day 29 are assumed to have no viral clearance.
Time Frame: Days 5, 7, 11, 14, 21, and 29 (saliva)
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 147 | 149
Participants
  Participants with Day 5 Samples who achieved sustained viral clearance: number analyzed (Participants) | 137 | 134
  Participants with Day 5 Samples who achieved sustained viral clearance | 21 | 9
  Participants with Day 7 Samples who achieved sustained viral clearance: number analyzed (Participants) | 135 | 131
  Participants with Day 7 Samples who achieved sustained viral clearance | 27 | 19
  Participants with Day 11 Samples who achieved sustained viral clearance: number analyzed (Participants) | 134 | 131
  Participants with Day 11 Samples who achieved sustained viral clearance | 55 | 40
  Participants with Day 14 Samples who achieved sustained viral clearance: number analyzed (Participants) | 134 | 128
  Participants with Day 14 Samples who achieved sustained viral clearance | 73 | 62
  Participants with Day 21 Samples who achieved sustained viral clearance: number analyzed (Participants) | 139 | 129
  Participants with Day 21 Samples who achieved sustained viral clearance | 98 | 83
  Participants with Day 29 Samples who achieved sustained viral clearance: number analyzed (Participants) | 136 | 130
  Participants with Day 29 Samples who achieved sustained viral clearance | 123 | 116
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; Test type: Superiority; p = 0.0227, Regression, Logistic — The p-value and risk difference reported was calculated based on the Day 5 timepoint; Risk Difference (RD) = 8.2, 95% CI 2-sided [1.15 to 15.31]

16. Secondary Outcome: SARS-CoV-2 Viral Load AUC Assessed by RT-qPCR From Saliva Samples
Description: The AUC from Day 1 through Day 29 was calculated according to the linear trapezoidal rule using the measured SARS-CoV-2 viral load above the lower limit of quantification. No AUC values will be calculated when Day 1 and/or Day 29 values are missing, or if there are more than 3 values missing in the profile.
Time Frame: Baseline to Day 29
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: log10 copies*day/mL
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 131 | 126
log10 copies*day/mL | 49.96 (36.54) | 57.60 (37.52)
Statistical Analysis 1: Comparison: ADG20 IM vs Placebo IM; Test type: Superiority; p = 0.1124, ANCOVA; Mean Difference (Final Values) = -6.93, 95% CI 2-sided [-15.49 to 1.64]

17. Secondary Outcome: Incidence of Treatment Emergent Adverse Events
Description: An AE is defined as any untoward medical occurrence in a participant enrolled into this study regardless of its causal relationship to the study drug. AEs occurring from when the participant signed the ICF until the Month 14 (EOS) visit or discontinuation from study was recorded
Time Frame: 14 months
Population: Percent of participants who reported at least one TEAE.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 192 | 200
Participants | 75 | 87

18. Secondary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Changes From Baseline in Clinical Laboratory Test (PCS Defined Per Statistical Analysis Plan)
Description: A PCS value is defined as any DAIDS grade 4 post-baseline or any increase of 2 or more DAIDS grades post-baseline, except for PCS low creatinine clearance, which is defined as any DAIDS Grade 4 post-baseline or any DAIDS grade shift from 0 to 3. Laboratory parameters not graded by DAIDs will be defined as PCS based on the criteria in the SAP (Appendix K.)
Time Frame: 14 Months
Population: Safety Set: All participants who received any amount of study drug. Participants were analyzed based on the actual treatment (ADG20 versus Placebo) received. Data presented for any analyte with >/= 2% in any arm.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 192 | 200
Participants
  Lymphocytes (10^9/L) - L | 3 | 4
  Alanine Aminotransferase (U/L) - H | 6 | 10
  Albumin (g/L) - L | 0 | 5
  Creatinine (mcmol/L) - H | 26 | 23
  Creatinine Clearance, Estimated (mL/min/1.73m2) - L | 15 | 18
  Glucose (mmol/L) - H | 12 | 16
  Sodium (mmol/L) - L | 1 | 4
  Urea Nitrogen (mmol/L) - H | 26 | 21
  Prothrombin Intl. Normalized Ratio - H | 5 | 1
  Prothrombin Time (sec) - H | 7 | 3

19. Secondary Outcome: Number of Participants With Potentially Clinically Significant (PCS) Changes From Baseline in Vital Sign Parameters (PCS Defined Per Statistical Analysis Plan)
Time Frame: 14 Months
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 192 | 200
participants
  SBP <=90 mmHg or Decrease >=20 mmHg | 17 | 23
  SBP >=180 mmHg or Increase >=20 mmHg | 29 | 26
  DBP <=50 mmHg or Decrease >=15 mmHg | 25 | 26
  DBP >=105 mmHg or Increase >=15 mmHg | 24 | 31
  HR <=50 bpm or Decrease >=15 bpm [a] | 78 | 96
  HR >120 bpm or Increase >=15 bpm | 20 | 25
  Temp <35 C or Decrease >=1 C [b] | 60 | 56
  Temp >=38 C or Increase >=1 C [c] | 5 | 17
  RR <=8 breaths/min or Decrease >=4 bpm | 20 | 25
  RR >=30 breaths/min or Increase >=10 bpm [d] | 2 | 2
  SpO2 <=93% or Decrease >=3% | 14 | 19

20. Secondary Outcome: Incidence of ADA to ADG20
Time Frame: 11 months
Population: All participants in the Safety Set who had a valid immunogenicity test result before the dose of study drug, and at least 1 valid result after the dose of study drug; analysis limited to participants who received ADG20 only.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 137 | 0
Participants | 12 | 0

21. Secondary Outcome: Genotypic Characterization of Viral Isolates for Reduced Susceptibility to ADG20 (G504 Mutations)
Description: Post-baseline Treatment-emergent Variations at Amino Acid Positions Associated with Reduced Susceptibility to ADG20 (>/= 15% Allele frequency); data limited to mutations observed.
Time Frame: Through Day 29
Population: Participants with any mutation at a monitored position >/= 15% allele frequency, in the population that had a qualifying (passed QC testing) baseline and post-baseline Whole Genome Sequencing sample.
Measure: Count of Participants; unit: Participants
Arm/Group | ADG20 IM | Placebo IM
Number analyzed (Participants) | 95 | 119
Participants | 3 | 0

ADVERSE EVENTS:
Time Frame: Baseline through Month 14
Description: safety analysis set
Arm/Group | ADG20 IM | Placebo IM
All-Cause Mortality (participants affected / at risk) | 2/192 | 7/200
Serious Adverse Events (participants affected / at risk) | 18/192 | 36/200
Other Adverse Events (participants affected / at risk) | 23/192 | 16/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADG20 IM (N=192) | Placebo IM (N=200)
COVID-19 pneumonia (Infections and infestations) | 8 | 24
Pneumonia bacterial (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Listeriosis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ADG20 IM (N=192) | Placebo IM (N=200)
Injection site pain (General disorders) | 23 | 16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04805671/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-03): https://cdn.clinicaltrials.gov/large-docs/71/NCT04805671/SAP_001.pdf